CLINICAL TRIAL: NCT07161570
Title: Effectiveness of Virtual Reality Digital Therapeutics for Seasonal Affective Disorder.
Brief Title: Virtual Reality Digital Therapeutics for Seasonal Affective Disorder
Acronym: VR-SAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Reneural Technologies Ltd. (Unknown); Aerial Icon Ltd. (Unknown); Innovate UK, UKRI (Unknown)
Responsible Party: Principal Investigator, Debora de Vasconcelos e Sa, Principal Investigator, Anglia Ruskin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10149188
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Seasonal Affective Disorder (SAD)
Keywords: SAD; VR
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) intervention (Experimental): 10-min VR intervention
  Interventions: Device: Virtual Reality (VR) Intervention
- Light Box (LB) intervention (Active Comparator): 30-min LB intervention
  Interventions: Device: Light Box (LB) intervention

INTERVENTIONS:
Device: Virtual Reality (VR) Intervention — 10-min VR intervention, once a day, everyday for 14 days.
  Arms: Virtual reality (VR) intervention
Device: Light Box (LB) intervention — 30-min LB intervention once a day, everyday for 14 days.
  Arms: Light Box (LB) intervention

SUMMARY:
Seasonal Affective Disorder (SAD) is commonly treated with bright light therapy. Virtual reality (VR) is an immersive computer-generated environment, which has been used to treat mental health difficulties, such as depression, social anxiety and stress. This study aims to compare the use of VR with bright light therapy in treating SAD.

Participants will be randomly allocated to either the VR condition or the light box condition and instructed to use the respective device every day for 14 days.

DETAILED DESCRIPTION:
Seasonal Affective Disorder (SAD) affects approximately 1 in 20 people in the UK during the winter months, with significant impacts on wellbeing and productivity. SAD is commonly treated with bright light treatment, alone or in combination with psychological therapy or antidepressants. Virtual reality (VR) is an immersive computer-generated environment. VR technology has been applied to treat a range of mental health conditions, including depression, anxiety, and stress. However, the possible contribution of this technology to the treatment of SAD has not been explored. This study aims to test the effectiveness of a VR intervention in alleviating symptoms of SAD compared to standard bright light treatment.

The investigators aim to recruit 60 participants who self-identify or have been diagnosed with SAD and who report moderate to severe symptoms. Participants are also required to be 18 years or older, a UK resident and able to access internet and attend the Anglia Ruskin University Cambridge campus. Participants will be excluded from the study if they declare suffering from epilepsy or having previously experienced adverse effects when using VR or light box devices. Participants will also be excluded if they are taking photosensitizing medications or have significant retinal pathology, or if they are currently receiving active treatment for SAD, including antidepressant medication, bright light treatment, or psychological treatment (such as Cognitive Behavioural Therapy). Recruitment will occur during the winter months, between November 2025 and March 2026.

After consenting, potential participants will be asked to complete some measures assessing their typical seasonal mood variation, to check eligibility to participate. If eligible, they will be asked to complete demographic questions and questionnaires measuring their current mood state and symptoms. Participants will then be randomly allocated to either the VR condition or the light box condition. Those allocated to the VR-condition, will be instructed to use the VR headset for 10 minutes within the first hour after waking, every day for 14 days. Those allocated to the light box intervention, will be instructed to use the light box for 30 minutes within the first hour after waking, every day for 14 days. Before and after each session, participants will be asked to record their current mood. At the end of the 14-day period, participants will return the headset or the light box and complete the final symptom and mood state questionnaires and questions regarding their experience. One week later, participants will be asked to complete a follow-up questionnaire about their mood and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English and capable of giving informed consent
* 18 or older
* resident in the United Kingdom and
* able to access internet and attend Anglia Ruskin University's Cambridge campus
* must self-identify or have been diagnosed with SAD, with moderate to severe symptoms

Exclusion Criteria:

* declared suffering from epilepsy (due to the risk that seizures may be triggered by VR use).
* currently using photosensitizing medications or have significant retinal pathology, due to potentially detrimental effects of light box use. For other ophthalmologic conditions, consultation with an ophthalmologist will be recommended.
* currently receiving active treatment for SAD, including antidepressant medication (less than 3 months), bright light treatment, or psychotherapy (e.g. CBT for seasonal affective disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in levels of mood and depressive symptoms | From baseline (day 1 to 7) to follow-up (day 28) of treatment
  Assessed by standardised psychological scales (Patient Health Questionnaire-9 (total score ranges from 0 to 27 with higher scores indication depression severity) and Positive and Negative Affect Schedule-Short Form (scores range from 10 to 50, with higher scores on the Positive Affect scale representing higher levels of positive affect, and higher scores on the Negative Affect scale representing higher levels of negative affect) and Visual Analogue Scales (0 to 100% with higher scores indicating better mood).

SECONDARY OUTCOMES:
Participant engagement, experience and satisfaction of the intervention | From baseline (day 1 to 7) to end of follow-up (day 28) treatment
  Assessed by self-report survey including written qualitative feedback (short online feedback form focusing on ease of use, perceived benefits and disadvantages), usage data (e.g., session attendance, frequency, duration, completion time) dropout rates and adverse effects reported.

CONTACTS AND LOCATIONS:
Overall Officials: Debora Vasconcelos e Sa, PhD, Principal Investigator — Anglia Ruskin University; Jane Scott, PhD, Study Director — Anglia Ruskin University

IPD SHARING:
Plan to Share IPD: Yes
This study will be written up to be published in peer-reviewed journals and anonymised data will be submitted to an online data repository (e.g., Figshare; Open Science Foundation).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon study completion December 2026.
Access Criteria: Findings from this study will be submitted for publication in peer-reviewed journals and anonymised findings will be included in an online data repository (e.g., Figshare; Open Science Foundation).